CLINICAL TRIAL: NCT00193206
Title: Phase II Trial of Dose Dense Neo-adjuvant Gemcitabine, Epirubicin, ABI-007 (GEA) in Locally Advanced or Inflammatory Breast Cancer
Brief Title: Neo-adjuvant Gemcitabine, Epirubicin, ABI-007 (GEA) in Locally Advanced or Inflammatory Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Eli Lilly and Company (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 73
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2012-11-30 (Estimated); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: Locally Advanced Breast Cancer; Inflammatory Breast Cancer; Breast Cancer; Abraxane; nab Paclitaxel; Epirubicin; Gemcitabine; Gemzar
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Gemcitabine; Epirubicin; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Patients were treated with 6 doses of neoadjuvant gemcitabine 2000 mg/m2, epirubicin 50 mg/m2, and albumin-bound paclitaxel 175 mg/m2 intravenously administered at 14-day intervals. Following neoadjuvant chemotherapy, patients underwent either mastectomy or breast conservation surgery; pathologic response to treatment was assessed. Postoperatively, patients received 4 doses of gemcitabine 2000 mg/m2 with albumin-bound paclitaxel 220 mg/m2 at 14-day intervals. Pegfilgrastim 6 mg was administered subcutaneously on day 2 following each dose of chemotherapy.
  Interventions: Drug: Gemcitabine; Drug: Epirubicin; Drug: Albumin-bound Paclitaxel

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 2000 mg/m2 IV D1 q 14 days x 6 cycles
  Other Names: Systemic therapy; Gemzar
Drug: Epirubicin — Epirubicin 50 mg/m2 D1 q 14 days x 6 cycles
  Other Names: Systemic therapy; Ellence
Drug: Albumin-bound Paclitaxel — ABI-007 175 mg/m2 D1 q 14 days x 6 cycles
  Other Names: Systemic therapy; ABI-007; Abraxane

SUMMARY:
In this trial we will evaluate ABI-007 with gemcitabine and epirubicin, utilizing the biweekly pegfilgrastim support, in order to further improve upon the effectiveness and favorable toxicity of this triplet.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be receive both induction neo-adjuvant regimen and a postoperative adjuvant regimen:

Induction Neo-adjuvant: Epirubicin + Gemcitabine + ABI-007 + Pegfilgrastim

Postoperative Adjuvant: Gemcitabine + ABI-007 + Pegfilgrastim

Upon completion of chemotherapy, all ER and/or PR+ patients will receive Tamoxifen or an aromatase inhibitor at physician discretion.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Locally advanced/inflammatory adenocarcinoma of the breast
* 18 years of age or older
* Normal heart function
* Able to perform activities of daily living with minimal assistance
* No prior chemotherapy for breast cancer
* Adequate bone marrow, liver and kidney function
* No evidence or history of significant cardiovascular abnormalities
* Sentinel node or axillary dissection
* Sign an informed consent form

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Pregnant or breast feeding
* History of heart disease with congestive heart failure
* Heart attack within the previous 6 months
* Prior chemotherapy or hormone therapy for breast cancer
* History of active uncontrolled infection

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2005-09; Primary Completion 2008-10 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Yardley, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (13):
- United States (13):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Hematology Oncology Life Center, Alexandria, Louisiana
  - Mercy Hospital, Portland, Maine
  - Oncology Hematology Care, Cincinnati, Ohio
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Chattanooga Oncology and Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Peninsula Cancer Institute, Newport News, Virginia

REFERENCES:
- [Background] Yardley DA, Zubkus J, Daniel B, Inhorn R, Lane CM, Vazquez ER, Naot Y, Burris HA 3rd, Hainsworth JD. A phase II trial of dose-dense neoadjuvant gemcitabine, epirubicin, and albumin-bound paclitaxel with pegfilgrastim in the treatment of patients with locally advanced breast cancer. Clin Breast Cancer. 2010 Oct 1;10(5):367-72. doi: 10.3816/CBC.2010.n.048. PMID 20670921

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Systemic Therapy
  ABI-007 : ABI-007 175 mg/m2 D1 q 14 days x 6 cycles
  Epirubicin : Epirubicin 50 mg/m2 D1 q 14 days x 6 cycles
  Gemcitabine : Gemcitabine 2000 mg/m2 IV D1 q 14 days x 6 cycles
Period: Preoperative Therapy
Arm/Group | Intervention
Started | 123
Completed | 116
Not Completed | 7
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — False Positive Pregnancy Test | 1
Period: Surgery
Arm/Group | Intervention
Started | 116
Completed | 116
Not Completed | 0
Period: Postoperative Therapy
Arm/Group | Intervention
Started | 116
Completed | 102
Not Completed | 14
Not completed — Withdrawal by Subject | 7
Not completed — Physician Decision | 3
Not completed — Intercurrent Illness | 2
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 123
Age, Continuous [Median (Full Range); unit: years] | 51 [29 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 123

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response
Description: For the purpose of this study, a pathologic complete response (pCR) was defined as no evidence of residual invasive tumor in the breast (pT0) and axillary lymph nodes (pN0), gross or microscopic, in the sample removed at the time of surgical resection. Residual ductal or lobular carcinoma in situ was not considered in pCR assessments. Percentage of participants who experienced pCR is reported.
Time Frame: 18 months
Population: 7 patients did not complete the study. Only the patients who had surgical procedures following neoadjuvant chemotherapy were included in the analysis as pathologic complete response is assessing the gross or microscopic response in the tissue sample resected at the time of surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 116
Participants | 23

2. Secondary Outcome: Clinical Response Rates
Description: Clinical response rate is defined as percentage of patients whose disease decreased (Partial response - PR) and/or disappeared (Complete response - CR) after treatment). Clinical tumor response was defined as complete if there was no clinical evidence of palpable tumor in either the breast or axilla at the time of surgery. Reduction of total tumor size >50 % at the time surgery was considered a clinical partial response. Evaluations are based on Response Evaluation Criteria in Solid Tumors (RECIST)
Time Frame: 18 months
Population: All patients who received neoadjuvant chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 123
Participants | 109

3. Secondary Outcome: Time to Disease Progression
Description: Time to progression is the length of time from the start of treatment until the disease progressed. Progressive disease is defined as an increase of >25% in the total calculated product of the tumor's measurements or development of a new lesion. Evaluations are based on Response Evaluation Criteria in Solid Tumors (RECIST)
Time Frame: 36 months
Measure: Median (Full Range); unit: months
Arm/Group | Intervention
Number analyzed (Participants) | 123
months | 13.7 [1.5 to 29.8]

4. Secondary Outcome: Rates of Breast Preservation
Description: Number of patients who underwent breast conservation after neo adjuvant chemotherapy
Time Frame: 18 months
Population: patients who had completed all 6 prescribed doses of neoadjuvant chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 116
Participants | 26

ADVERSE EVENTS:
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 22/123
Other Adverse Events (participants affected / at risk) | 41/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=123)
Cardiac Ischemia/Infarction (Cardiac disorders) | 1 (1) — Angina
Infection - Skin (Infections and infestations) | 3 (3) — Cellulitis
Pain - Chest (Cardiac disorders) | 2 (2)
Infection - Gastrointestinal (Infections and infestations) | 1 (1) — Colitis
Dehydration (Gastrointestinal disorders) | 2 (2)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2 (2)
Infection - Vein (Infections and infestations) | 2 (2) — Septic Thrombophlebitis
Death (General disorders) | 1 (1) — Intercurrent Illness
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - Liver (Hepatobiliary disorders) | 1 (1)
Infection - Pneumonia (Infections and infestations) | 1 (1)
Infection - Skin (Infections and infestations) | 3 (4) — Port Site Infection
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Progressive Disease
Neurology - Other (Psychiatric disorders) | 1 (1) — Suicidal Ideations
Weakness (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=123)
Neutrophils (Blood and lymphatic system disorders) | 13 — Neutropenia
Platelets (Blood and lymphatic system disorders) | 7 — Thrombocytopenia
Arthralgia/Myalgia (Musculoskeletal and connective tissue disorders) | 8
Fatigue (General disorders) | 7
Thrombosis/Thrombus/Embolism (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.